CLINICAL TRIAL: NCT05996406
Title: Venetoclax Combined with Dexamethasone for Newly Diagnosed Light-Chain Amyloidosis Patients with Translocation (11;14): a Multicenter Phase 2 Study
Brief Title: Venetoclax and Dexamethasone for Newly Diagnosed Light-Chain Amyloidosis with Translocation (11;14)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Jian Li, Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ven-D001
Record Dates: First submitted 2023-08-09; First posted 2023-08-18 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Light Chain (AL) Amyloidosis; CCND1 Translocation; Venetoclax
MeSH Terms: conditions — Amyloidosis | interventions — venetoclax; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ven-D (Experimental): Venetoclax combined with dexamethasone
  Interventions: Drug: Venetoclax; Drug: Dexamethasone Oral

INTERVENTIONS:
Drug: Venetoclax — Venetoclax 400mg po qd for 1 year
Drug: Dexamethasone Oral — Dexamethasone 40mg po qw for the first 6 months, then 10mg po qw for the next 6 months

SUMMARY:
Venetoclax is considered as a promising agent for light-chain (AL) amyloidosis due to the high percentage of t(11;14). Several retrospective studies showed venetoclax-based therapy could induce rapid and profound hematologic response in AL patients with favorable safety profile. As an oral agent with encouraging data, it is worth to prospectively evaluate the efficacy and safety of venetoclax in untreated AL amyloidosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proved treatment-naïve AL amyloidosis
* Fluorescence in situ hybridization (FISH) t(11;14) ≥ 10%
* dFLC > 50mg/L

Exclusion Criteria:

* Co-morbidity of uncontrolled infection
* Co-morbidity of other active malignancy
* Co-diagnosis of multiple myeloma or waldenstrom macroglobulinemia
* Co-morbidity of grade 2 Mobitz II or grade 3 atrioventricular block (expect for those with implanted pacemaker)
* Co-morbidity of sustained or recurrent nonsustained ventricular tachycardia
* Seropositive for human immunodeficiency virus
* Hepatitis B virus (HBV)-DNA > 1000 copies/mL
* Seropositive for hepatitis C (except in the setting of a sustained virologic response)
* Systemic treatment with moderate or strong cytochrome P450 3A （CYP3A） inducers, moderate or strong CYP3A inhibitors within 7 days prior to the first dose of study drug
* Neutrophil <1×10E9/L，hemoglobin < 8g/dL，or platelet < 100×10E9/L.
* Severely compromised hepatic or renal function: alanine transaminase (ALT) or aspertate aminotransferase (AST) > 2.5 × upper limit of normal (ULN), total bilirubin > 3 × ULN，eGFR < 15 mL/min, or receiving renal replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR)+very good partial response (VGPR) at 3 months after treatment initiation | 3 months after treatment initiation

SECONDARY OUTCOMES:
Overall survival | 2 years
Time to next treatment | 2 years
CR+VGPR at 1 month after treatment initiation | 1 month after treatment initiation
CR+VGPR at 6 months after treatment initiation | 6 months after treatment initiation
CR+VGPR at 12 months after treatment initiation | 12 months after treatment initiation
Difference between involved and uninvolved free light chain (dFLC) < 10mg/L | at 1, 3, 6 and 12 months after treatment initiation
Involved free light chain (iFLC) ≤ 20mg/L | at 1, 3, 6 and 12 months after treatment initiation
Minimal residual disease (MRD) negativity | 12 and 24 months after treatment initiation
Time to hematologic response | 1 year
Time to hematologic CR | 1 year
Cardiac response | at 3, 6, 12 and 24 months after treatment initiation
Renal response | at 3, 6, 12 and 24 months after treatment initiation
Hepatic response | at 3, 6, 12 and 24 months after treatment initiation
Time to cardiac response | 2 years
Time to renal response | 2 years
Time to hepatic response | 2 years
Adverse events | treatment initiation to 30 days after last dose of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China